CLINICAL TRIAL: NCT00764413
Title: Treatment With Methylprednisolone in Acute Exacerbations of Multiple Sclerosis: Enhanced Effect With Nighttime Treatment?
Brief Title: Chronotherapy in Acute Multiple Sclerosis (MS) Attack
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low inclusion frequency and not enough human resources for completing study
Sponsor: Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15002; 150134 (Other Grant/Funding Number: Innlandet Hospital Trust); 2008-002025-37 (EudraCT Number)
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-02

CONDITIONS: Multiple Sclerosis
Keywords: EDSS; methylprednisolone; circadian rhythms; MSFC
MeSH Terms: conditions — Multiple Sclerosis | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Both study arms receive both active treatment = methylprednisolone and an inactive treatment = Sodium chlorid (dummy)
  Interventions: Drug: methylprednisolone; Drug: Sodium chlorid
- 2 (Active Comparator): Both arms receives both active treatment and inactive treatment = dummy. Active treatment is methylprednisolone, inactive treatment is sodium chlorid.
  Interventions: Drug: methylprednisolone; Drug: Sodium chlorid

INTERVENTIONS:
Drug: methylprednisolone — 1 gram intravenous a day for 3 days
  Other Names: Solu-Medrol. ACT-nr:H02A B04
Drug: Sodium chlorid — Sodium chlorid 9mg/ml 500 ml per day in 3 days
  Other Names: ATC: B05B B01

SUMMARY:
The Immunological system is showing a diurnal rhythmicity. The Mediators that enhances inflammation are at highest level during the night. At the same time the endogenous production of cortisol is at its lowest. We want to study if there is a better effect of treatment with Methylprednisolone for acute MS-attacks if given at nighttime. The effect will be measured in relation to neurological deficits and function with Kurtzkes Expanded Disability Status Score (EDSS) and Multiple Sclerosis Functional Composite (MSFC). We want to see if the mean improvement in EDSS is greater in the group receiving treatment at night opposed to the group that get treatment during the daytime.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing remitting MS
* EDSS-score before the actual attack < 6.0
* Acute MS-attack with indication for treatment with steroids
* Symptoms >24 hours < 4 weeks
* Age 18 years or older

Exclusion Criteria:

* Prior enrollment in this study
* Ongoing serious infection that is a contraindication for treatment with steroids
* Pregnancy
* Medical situations (prior acute diseases) where treatment with intravenous steroids over short period of time is contraindicated or not favorable.
* Enhanced cognitive dysfunction
* Treatment with p.o or i.v steroids within 3 weeks prior to date of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The difference in mean changes in EDSS-score between the group receiving treatment during the night opposed to during the day. | At admittion, directly after treatment, ca 30 days after treatment

SECONDARY OUTCOMES:
The difference in MSFC-score in the two groups | At admittion, directly after treatment, ca 30 days after treatment
Side effect registered by the patient | At admittion (baseline), during treatment, directly after treatment
The patient's quality of life | At admittion, directly after treatment, 7 days and ca 30 days after treatment
MRI - volume and number for MS-lesions, Gd-enhancement | At admission, directly after treatment and ca 30 days after treatment
Fatigue | Before, after and ca 30 days after treatment
Depression | Before, after and ca 30 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anette H Farmen, Physician/MD, Study Director — Innlandet Hospital Trust Lillehammer, Neurological Department; Kristin I Løken-Amsrud, Physician/MD, Study Director — Innlandet Hospital Trust Lillehammer, Neurological Department; Elisabeth G Celius, MD/PhD, Study Chair — Oslo University Hospital, Ullevål, Neurological Department; Per O Vandvik, MD/PhD, Study Chair — Innlandet Hospital Trust Gjøvik, Department of Internal medicin; Trygve Holmøy, MD/PhD, Study Chair — Oslo University Hospital, Ullevål, Neurological department
Locations (1):
- Innlandet Hosptal Trust-Lillehammer, Neurological Department, Lillehammer, Oppland, Norway